CLINICAL TRIAL: NCT02738138
Title: A Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Adults With Chronic Hepatitis C Virus (HCV) Genotype 1 - 6 Infection and Human Immunodeficiency Virus-1 (HIV-1) Co-Infection (EXPEDITION-2)
Brief Title: A Study to Evaluate the Efficacy and Safety of Experimental Drugs ABT- 493/ABT-530 in Adults With Chronic Hepatitis C Virus Genotype 1-6 Infection and Human Immunodeficiency Virus -1 Coinfection (EXPEDITION-2)
Acronym: EXPEDITION-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-730; 2015-005577-20 (EudraCT Number)
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C Virus Infection; Human Immunodeficiency Virus Infection; Chronic Hepatitis C; Compensated Cirrhosis and Non-cirrhotics
Keywords: HCV Genotype 3; Non-cirrhotic; HCV Genotype 1; HCV Genotype 6; Human Immunodeficiency Virus (HIV) Infection; HCV Genotype 5; HCV Treatment Naive; HCV Genotype 4; HCV Treatment Experienced; HCV Genotype 2; Hepatitis C Virus (HCV) Infection; Compensated Cirrhosis
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic; Infections | interventions — pibrentasvir; glecaprevir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABT-493/ABT-530 for 8 weeks (Experimental): HCV Genotype (GT)1-6/HIV-1 co-infected non-cirrhotic subjects treated with ABT-493/ABT-530 300 mg/120 mg once a day (QD) for 8 weeks
  Interventions: Drug: ABT-493 coformulated with ABT-530
- ABT-493/ABT-530 for 12 weeks (Experimental): HCV GT1-6/HIV-1 co-infected subjects with compensated cirrhosis treated with ABT-493/ABT-530 300 mg/120 mg once a day (QD) for 12 weeks
  Interventions: Drug: ABT-493 coformulated with ABT-530

INTERVENTIONS:
Drug: ABT-493 coformulated with ABT-530 — Tablet
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; MAVYRET

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ABT-493/ABT-530 in adults with chronic hepatitis C virus genotype 1-6 infection and human immunodeficiency virus-1 co-infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age at time of Screening.
2. Screening laboratory result indicating Hepatitis C virus (HCV) genotype (GT)1-, 2-, 3-, 4-, 5-, or 6-infection.
3. Subject has positive anti-HCV antibody (Ab) and plasma HCV ribonucleic acid (RNA) viral load greater than or equal to 1000 IU/mL at Screening visit.
4. Subjects must be HCV treatment-naïve (i.e., subject has never received a single dose of any approved or investigational anti-HCV medication) or HCV treatment-experienced (subject who has failed prior IFN or pegylated-interferon [pegIFN] with or without ribavirin [RBV], or sofosbuvir [SOF] plus RBV with or without pegIFN). GT3 subjects must be HCV treatment-naïve. Previous HCV treatment must have been completed greater than or equal to 2 months prior to Screening.
5. Subjects naïve to antiretroviral treatment (ART) must have CD4+ count greater than or equal to 500 cells/mm^3 (or CD4+ % greater than or equal to 29%) at Screening; or Subjects on a stable ART regimen must have

   * CD4+ count greater than or equal to 200 cells/mm^3 (or CD4+ % greater than or equal to 14%) at Screening; and
   * Plasma HIV-1 RNA below lower limit of quantification (LLOQ) at Screening and at least once during the 12 months prior to Screening.

Exclusion Criteria:

1. Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
2. Positive test result at Screening for hepatitis B surface antigen (HBsAg).
3. Positive Human Immunodeficiency virus, type 2 (HIV-2) Ab at Screening.
4. Receipt of any other investigational or commercially available direct acting anti-HCV agents other than sofosbuvir (e.g., telaprevir, boceprevir, simeprevir, paritaprevir, grazoprevir, daclatasvir, ledipasvir, ombitasvir, elbasvir or dasabuvir).
5. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive ABT-493/ABT-530.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Background] Rockstroh JK, Lacombe K, Viani RM, Orkin C, Wyles D, Luetkemeyer AF, Soto-Malave R, Flisiak R, Bhagani S, Sherman KE, Shimonova T, Ruane P, Sasadeusz J, Slim J, Zhang Z, Samanta S, Ng TI, Gulati A, Kosloski MP, Shulman NS, Trinh R, Sulkowski M. Efficacy and Safety of Glecaprevir/Pibrentasvir in Patients Coinfected With Hepatitis C Virus and Human Immunodeficiency Virus Type 1: The EXPEDITION-2 Study. Clin Infect Dis. 2018 Sep 14;67(7):1010-1017. doi: 10.1093/cid/ciy220. PMID 29566246
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Naganuma A, Chayama K, Notsumata K, Gane E, Foster GR, Wyles D, Kwo P, Crown E, Bhagat A, Mensa FJ, Otani T, Larsen L, Burroughs M, Kumada H. Integrated analysis of 8-week glecaprevir/pibrentasvir in Japanese and overseas patients without cirrhosis and with hepatitis C virus genotype 1 or 2 infection. J Gastroenterol. 2019 Aug;54(8):752-761. doi: 10.1007/s00535-019-01569-7. Epub 2019 Mar 13. PMID 30868245
- [Derived] Foster GR, Dore GJ, Wang S, Grebely J, Sherman KE, Baumgarten A, Conway B, Jackson D, Asselah T, Gschwantler M, Tomasiewicz K, Aguilar H, Asatryan A, Hu Y, Mensa FJ. Glecaprevir/pibrentasvir in patients with chronic HCV and recent drug use: An integrated analysis of 7 phase III studies. Drug Alcohol Depend. 2019 Jan 1;194:487-494. doi: 10.1016/j.drugalcdep.2018.11.007. Epub 2018 Nov 24. PMID 30529905
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 35-day screening period.
Groups:
- ABT-493/ABT-530 for 8 Weeks: HCV GT1-6/HIV-1 co-infected non-cirrhotic subjects treated with ABT-493/ABT-530 300 mg/120 mg once a day (QD) for 8 weeks
Period: Overall Study
Arm/Group | ABT-493/ABT-530 for 8 Weeks | ABT-493/ABT-530 for 12 Weeks
Started | 137 | 16
Completed | 134 | 15
Not Completed | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other - not further specified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-493/ABT-530 for 8 Weeks | ABT-493/ABT-530 for 12 Weeks | Total
Number analyzed (Participants) | 137 | 16 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.00 (10.22) | 50.00 (8.36) | 45.00 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 1 | 25
  Male | 113 | 15 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 1 | 25
  White | 106 | 15 | 121
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of active study drug.
Time Frame: 12 weeks after last dose of study drug
Population: Per protocol, all efficacy analyses were performed using the intention-to-treat (ITT) population (all enrolled participants who received at least 1 dose of study drug); in addition, efficacy analyses were performed overall, combining Treatment Arms A and B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ABT-493/ABT-530: HCV GT1-6/HIV-1 co-infected participants treated with ABT-493/ABT-530 300 mg/120 mg once a day (QD)
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 153
percentage of participants | 98.0 [95.8 to 100.0]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Up to 12 weeks
Population: Per protocol, all efficacy analyses were performed using the ITT population; in addition, efficacy analyses were performed overall, combining Treatment Arms A and B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 153
percentage of participants | 0.7 [0.1 to 3.6]

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: Per protocol, all efficacy analyses were performed using the ITT population including only those participants who had post-treatment data available, excluding reinfection (N = 151). In addition, efficacy analyses were performed overall, combining Treatment Arms A and B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-493/ABT-530
Number analyzed (Participants) | 151
percentage of participants | 0 [0.0 to 2.5]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and SAEs are defined as any AE or SAE from the first dose of study drug to 30 days after the last dose of study drug (up to 16 weeks).
Groups:
- ABT-493/ABT-530 for 8 Weeks: HCV GT1-6/HIV-1 co-infected non-cirrhotic subjects will be treated with ABT-493/ABT-530 300 mg/120 mg once a day (QD) for 8 weeks
- ABT-493/ABT-530 for 12 Weeks: HCV GT1-6/HIV-1 co-infected subjects with compensated cirrhosis will be treated with ABT-493/ABT-530 300 mg/120 mg once a day (QD) for 12 weeks
Arm/Group | ABT-493/ABT-530 for 8 Weeks | ABT-493/ABT-530 for 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/16
Serious Adverse Events (participants affected / at risk) | 3/137 | 1/16
Other Adverse Events (participants affected / at risk) | 50/137 | 7/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-493/ABT-530 for 8 Weeks (N=137) | ABT-493/ABT-530 for 12 Weeks (N=16)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
CALCULUS URINARY (Renal and urinary disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-493/ABT-530 for 8 Weeks (N=137) | ABT-493/ABT-530 for 12 Weeks (N=16)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL SOUNDS ABNORMAL (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 12 (12) | 1 (1)
FATIGUE (General disorders) | 18 (18) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 1 (1)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 (12) | 0 (0)
DIZZINESS (Nervous system disorders) | 3 (3) | 1 (1)
HEADACHE (Nervous system disorders) | 12 (12) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (2) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-07-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT02738138/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT02738138/SAP_001.pdf